CLINICAL TRIAL: NCT02823756
Title: The Short-Term Effects of Manipulation and Physical Therapy on Physical Activity Levels
Brief Title: Short-Term Effects of PT on Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Wayne Brewer, Assistant Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17852
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Low Back Pain; Motor Activity; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Motor Activity; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Therapy (Experimental): Treatment arm: manipulation, exercise, and education
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Physical Therapy — Exercise, education, spinal manipulation

SUMMARY:
The primary purpose is to examine the impact that physical therapy (PT) interventions, including manipulations, have on physical activity levels outside of the clinical environment in persons with low back pain (LBP) as measured both objectively with an accelerometer and subjectively with questionnaires.

The secondary purpose is to determine if a relationship exists between objective physical activity, self-perceived disability pain catastrophizing thoughts, BMI, age, six-minute walk distance, lower extremity muscle endurance.

The tertiary purpose is to assess the predictive value that a standing manual lumbar unloading technique has for relief of pain following manipulation

DETAILED DESCRIPTION:
At session 1: Participants are screened for eligibility. Baseline outcome measures are conducted (self-report questionnaires and physical performance tests). Accelerometer which is an instrument to measure physical activity is issued.

At session 2 (To occur at least one-week later): Accelerometer data is retrieved and downloaded to a computer. Participant numerically rates low back pain level at rest and in most painful position. Participant receives a manual distraction procedure. Participant rates pain level again. Participant starts the physical therapy intervention (manipulation of the spine, muscular strengthening and cardiovascular exercise, education). Accelerometer is reissued again.

At session 3 (At least one-week later): Accelerometer is collected and data is retrieved. Participant continues with the intervention (manipulation, exercise, education).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient referred to outpatient PT with a LBP related diagnosis

  2. LBP without radiating pain distally to the knee > 3 months in duration

  3. Ability to read and write in English or Spanish

  4. Age between 18 and 70 years

  5. Able to ambulate independently without assistive devices

  6. Access to a computer or cell phone with an email address and/or the ability to receive short text messages

Exclusion Criteria:

* 1. No previous diagnosis, radiological evidence, or clinical signs and symptoms of instability, spondylolysis, spondylolisthesis, fracture, tumor or metastases to the spine

  2. No clinical indication of nerve root pathology such as: straight leg raise less than 45 degrees, asymmetric lower extremity deep tendon reflexes, lower extremity muscle strength deficits or radiating pain, numbness or tingling below the knee

  3. No surgical or biological fusion to the spine

  4. No previous spinal surgery

  5. No known diagnosis of osteoporosis or rheumatoid arthritis

  6. No use of oral steroids within the past 6 months

  7. No epidural injection over the previous 4-weeks to the lumbar spine region

  8. No current litigation, workman's compensation or disability claim for a low back injury

  9. No known pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity Levels | 2 weeks
  Accelerometer issued to subject at the initial data collection session and then data collected and downloaded one week later. Subject receives the intervention session, then is reissued the accelerometer. Subject returns the accelerometer one week after this intervention session with data that reflects physical activity levels that are after the intervention session

OTHER OUTCOMES:
Visual Analog Scale | 1 day
  A 10 cm horizontal line that the subject will use to descibe how intense their pain is before and after receiving a spinal manipulation by placing a vertical hash mark along the horizontal line to denote how intense his or her pain is.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne A Brewer, PhD, Principal Investigator — Texas Woman's University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer W, Swanson BT, Roddey TS, Adewale H, Ashmore C, Frerich J, Perrin C, Ortiz A. A pilot study to determine the effect of one physical therapy session on physical activity levels for individuals with chronic low back pain. BMC Res Notes. 2017 Dec 6;10(1):691. doi: 10.1186/s13104-017-3006-x. PMID 29208007